CLINICAL TRIAL: NCT01457287
Title: Cognitive Function and Fatigue in Cancer Patients After Chemotherapy: A Longitudinal Controlled Study in Patients With Colorectal Cancer
Brief Title: A Longitudinal Investigation of Cognitive Function in Colorectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Ian Tannock, UHN
Other Study IDs: COIT10
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, longitudinal, controlled study of cognitive function and fatigue in patients with apparently localized CRC treated with adjuvant or neoadjuvant chemotherapy. In addition to following each patient over time (i.e. acting as their own control), a separate control group will consist of patients with early stage CRC (Stage A or B) who have had surgical resection of their tumour, but who do not require adjuvant chemotherapy, or patients with stage C CRC who have declined chemotherapy.

Also included is a smaller sub-study of patients with limited metastatic CRC who are treated with more toxic chemotherapy

To compare changes in cognitive function, as compared to baseline assessment, of patients with CRC who do, or do not, receive 5FU-based chemotherapy. The primary measures of cognitive function are the High Sensitivity Cognitive Screen (HSCS) & Coghealth™.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years old
* Performance Status (PS) of 0-1 on the ECOG Performance Scale
* Life expectancy of at least 12 months
* Full recovery from any post operative sequelae
* Adequate hepatic function as documented by a serum bilirubin < 18umol/L, and LFTs within 1.5X normal range
* Patients with histologically confirmed, stage B or C colorectal cancer (CRC), who have undergone surgical resection and are about to commence chemotherapy.
* Patients due to receive neoadjuvant chemotherapy prior to surgery are also eligible.

Exclusion Criteria:

* Any major pre-existing psychiatric history or dementia, alcohol abuse, or currently using a psychotropic medication that might lead to cognitive problems, other than short acting benzodiazepines for nausea or sleep
* Any evidence of metastatic disease. If there is clinical suspicion of CNS involvement patients must have brain imaging (MRI or CT scan) prior to recruitment.
* Ongoing sepsis or uncontrolled infection, including HIV infection
* Pre-existing neurological condition likely to interfere with ability to perform cognitive testing
* Any other severe co-morbidity which, in the judgement of the investigator, would make the patient inappropriate for entry into this study
* Active cancer within the last 5 years other than squamous or basal cell carcinoma of the skin or cervical cancer in situ (except for CRC)
* Previous history of chemotherapy
* Minimal English skills such that subjects would be unable to follow simple, written English instructions and to read questionnaires of a grade 8 standard with the help of a research assistant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients being treated for Colorectal cancer at participating centres
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2003-10

PRIMARY OUTCOMES:
Cognitive Function | 2 years
  To compare changes in cognitive function, as compared to baseline assessment, of patients with CRC who do, or do not, receive 5FU-based chemotherapy. The primary measures of cognitive function are the High Sensitivity Cognitive Screen (HSCS) & Coghealth™.

SECONDARY OUTCOMES:
Potential mechanisms leading to fatigue and/or cognitive decline | 2 Years
  To evaluate potential mechanisms leading to fatigue and/or cognitive decline. To measure hemoglobin, serum levels of sex hormones (LH, FSH, estradiol (in women), testosterone (in men)), selected cytokines (TNF-α, IL-1 & IL-6), homocysteine, markers of blood coagulation (thrombin-anti-thrombin (TAT), prothrombin fragment 1 & 2, and d-dimers), and the apolipoprotein E genotype

CONTACTS AND LOCATIONS:
Overall Officials: Ian F Tannock, MD, PhD, DSc, Principal Investigator — UHN/PMH